CLINICAL TRIAL: NCT04548258
Title: Bone Changes Assessment in Screw-Retained Maxillary Implant Supported Complete Denture With Electric Welded Metal Framework Versus Cast One (Randomized Control,Split Mouth Trial)
Brief Title: Bone Changes Assessment in Screw-Retained Maxillary Complete Denture With Electric Welded Framework Versus Cast One
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Magdy Abd Elhakm Mohmed, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6420
Record Dates: First submitted 2020-08-28; First posted 2020-09-14 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Bone Resorption
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electric welded metal framework (Experimental): using electric welding device to intraorally join metal framework where the study aim to save time and cost and eliminate lab errors
  Interventions: Device: electric intraoral weilding
- conventional cast metal technique (Experimental): using the conventional casting technique to join metal framework and compare it with the electric welding technique
  Interventions: Device: casting

INTERVENTIONS:
Device: electric intraoral weilding — weilding metal framework to the implants in completely edentulous maxilla using electric weilding device intraorally
  Arms: electric welded metal framework
Device: casting — casting metal framework
  Arms: conventional cast metal technique

SUMMARY:
comparing bony changes around implants that will be joined by ametal framework either with electric weiling or with the conventional casting metal

DETAILED DESCRIPTION:
joining multiple implants together in the edentulous arches is considered agood solution, using the conventional casting technique has many disadvantages due to lab errors and time and cost consuming on ,the other hand the study aims to owercome these disadvantages using electric welding metal framework.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 30 to 65 years old.
* Absence of any medical disorder that could complicate the Surgical phase or affect osseointegration.
* The patients must be completely edentulous.
* The patient must have enough bone height for implants minimum length of 10mm and a minimum diameter of 5 mm.
* Patients with good oral hygiene.
* Complete denture wearer.
* Adequate inter arch space for screw retained prosthesis.
* Absence of any intra-oral pathological condition.

Exclusion Criteria:

Patients with recent extraction(less than three months).

* Patients with inflamed ridge or candida infection.
* Patients with flappyridge.
* Parafunctional habits.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
bony changes assessment | 12 months
  assessment of bone height changes around implants using digital periapical paralling imaging technique and the unit will be meagured in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University ,Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No